CLINICAL TRIAL: NCT04631328
Title: Sesame Street Growing Together Evaluation: Randomized Controlled Trial of a Professional Development Course for Early Care and Education Teachers
Brief Title: Sesame Street Growing Together Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Management Corporation (Other)
Collaborators: Sesame Workshop (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1903
Record Dates: First submitted 2020-07-22; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Family Engagement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Growing Together program
  Interventions: Other: Growing Together
- Control (No Intervention)

INTERVENTIONS:
Other: Growing Together — Growing Together is a suite of free, online research-informed professional development modules to help early childhood educators promote deeper family engagement and enrich teacher-parent interactions.
  Arms: Intervention

SUMMARY:
This study aims to evaluate the appeal and effectiveness of Sesame Workshop's Growing Together online professional development course.

ELIGIBILITY:
Inclusion Criteria:

Teachers:

* Work in an eligible center with a director who has agreed for the center to participate in the study
* Serve as the lead teacher in a classroom with at least 3 four year olds (can be a co-teacher and can teach a mixed age class)
* Have access to reliable, high-speed internet
* Have an email address that can be shared with researchers
* Read English enough to understand course materials and/or surveys
* Not have previously accessed the Growing Together course
* Be available during the timeframe of the study

Parents:

* Have a child who is 4 years old or about to be 4 years old during the weeks of the course enrolled in a classroom at least 3 days in a typical week with a teacher interested in participating in the study
* Have access to reliable, high-speed internet
* Have an email address that can be shared with researchers
* Read English enough to understand course materials and/or surveys
* Be available during the timeframe of the study

Exclusion Criteria:

Teachers:

* Working in an ineligible center
* Working in a center with a director who has not agreed for the center to participate in the study
* Not being a lead teacher
* Not teaching at least 3 four year olds
* Not having access to reliable, high-speed internet
* Not willing to share an email address with researchers
* Being unable to read English enough to understand course materials and/or surveys
* Having previously accessed the Growing Together course
* Not being available during the timeframe of the study

Parents:

* Not having a child who is 4 years old or about to be 4 years old during the weeks of the course
* Not having a child enrolled in a classroom at least 3 days in a typical week
* Not having a child enrolled in a classroom with a teacher interested in participating in the study
* Not having access to reliable, high-speed internet
* Not willing to share an email address with researchers
* Being unable to read English enough to understand course materials and/or surveys
* Not being available during the timeframe of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Family and Provider/Teacher Relationship Quality (FTPRQ) | Up to 12 weeks
  Self-report measure (teachers and parents) of the quality of family and teacher relationships.
Teachers' Sense of Efficacy Scale | Up to 12 weeks
  Teachers' self-efficacy in three areas: student engagement, instructional strategies, and classroom management.
Family Involvement Questionnaire (FIQ) | Up to 12 weeks
  Multi-dimensional parent-report scale of family involvement in early childhood education, reflecting levels of involvement of parent activity across home and classroom contexts.
Activities with Your Child | Up to 12 weeks
  Parent report of the frequency with which they or someone in their family engaged in a variety of activities with their child; adapted from the Head Start FACES studies parent interviews.

SECONDARY OUTCOMES:
Devereux Early Childhood Assessment for Preschoolers, Second Edition (DECA-P2) | Up to 12 weeks
  Behavior rating scale completed by parents and teachers. Provides an assessment of within-child protective factors related to resilience and a screener for behavioral concerns in children ages 3 through 5.

CONTACTS AND LOCATIONS:
Locations (1):
- PHMC, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT04631328/ICF_000.pdf